CLINICAL TRIAL: NCT01886508
Title: A Multicentre Trial of Nerve-Spring Radical Hysterectomy vs. Radical Hysterectomy for Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Tumor Hospital of Xin Jiang Medical University,China (Unknown); Gui Yang Maternal and Child Health Hospital,China (Unknown); The 152nd Hospital of chinese People's Liberation Army (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCT00270426
Record Dates: First submitted 2012-09-25; First posted 2013-06-26 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NSRH (Experimental): patients in Arm NSRH undergo nerve-spring radical hysterectomy (NSRH)
  Interventions: Procedure: Nerve-spring radical hysterectomy
- RH (Active Comparator): patients in Arm RH undergo radical hysterectomy (RH)
  Interventions: Procedure: radical hysterectomy

INTERVENTIONS:
Procedure: Nerve-spring radical hysterectomy — Nerve-spring radical hysterectomy that is reserve some pelvic autonomic nerves during radical hysterectomy. Reserve hypogastric nerve trunk during dissecting cardinal ligament. Reserve pelvic splanchnic nerve trunk during exsecting uterosacral ligament. Reserve bladder nerve of pelvic plexus during dissecting vesicouterine ligament.
  Arms: NSRH
Procedure: radical hysterectomy — Radical hysterectomy is Piver III hysterectomy and Q-M classification Type C1 hysterectomy.
  Arms: RH

SUMMARY:
The investigators designed this multicentre randomized study to investigate the clinical benefits of nerve-spring radical hysterectomy for cervical cancer. Patients with FIGO stage Ia2, Ib1, IIa1 and FIGO stage Ib2, IIa2 after neoadjuvant chemotherapy are randomized to either nerve-spring radical hysterectomy or radical hysterectomy. The primary endpoint are urodynamic outcome including maximum flow rate, residual volume, maximum vesical compliace, cystomctric capacity at first desire, and maximum cystomctric capacity. A total 240 patients (120 per treatment arm) are planned to accrue for this study within 7 years.

ELIGIBILITY:
Inclusion Criteria:

1. FIGO(2009) stage Ia2, Ib1, and IIa1 Untreated cervical cancer OR FIGO(2009) stage Ib2 and IIa2 cervical cancer that possible to surgery after neoadjuvant chemotherapy
2. Possible to radical hysterectomy or nerve-spring radical hysterectomy
3. Age: 17 to 60 years
4. No complication during operation
5. Written informed consent

Exclusion Criteria:

1. patients who underwent radiotherapy
2. Pathologically diagnosed Pathologically diagnosed squamous carcinoma, Small Cell Carcinoma, Small Cell Carcinoma
3. Patients who have uncontrolled diabetes or uncontrolled hypertension
4. patients with neurogenic bladder dysfunction
5. patients with uterine prolapse
6. Patients with psychiatric illness
7. Patients who have active infection
8. Patients who have had heart failure, unstable angina, or myocardial infarction within the past 6 months
9. Patients who are unable to undergo radical hysterectomy for complication of excessive obesity, liver cirrhosis, or bleeding tendency

Ages: 17 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
maximum flow rate measured by Urodynamic at 6 months postoperative | on 6 months postoperative
residual volume measured by Urodynamic at 6 months postoperative | on 6 months postoperative
maximum vesical compliace measured by Urodynamic at 6 months postoperative | on 6 months postoperative
cystometric capacity at first desire measured by Urodynamic at 6 months postoperative | on 6 months postoperative
maximum cystometric capacity (MCC) measured by Urodynamic at 6 months postoperative | on 6 months postoperative

SECONDARY OUTCOMES:
Time (days) to residual urine volume less than 100ml postoperative | from operation to residual urine volume less than 100ml, assessed up to 30 days
time (hours) to break wind postoperative | from operation to have the first break wind, assessed up to 72 hours
time (hours) to defecation postoperative | from operation to have the first defection, assessed up to 72 hours
Number of participants with adverse events | From date of operation until the date of first documented adverse event or date of death from any cause, whichever came first, assessed up to 5 years
Score of MHU rating scales at 6 months postoperative | on 6 months postoperative
overall survival | From date of operation until the date of death from any cause, assessed up to 5 years
progression-free survival | From date of operation until the date of relapse or date of death from any cause, whichever came first, assessed up to 5 years
Score of C-30 life quality rating scales at 6 months postoperative | on 6 months postoperative
Score of CX-24 life quality rating scales at 6 months postoperative | on 6 months postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical University, China, Guangzhou, Guangdong, China